CLINICAL TRIAL: NCT01861483
Title: Resection and Reconstruction of Major Vessels in Biliary Tract Cancers
Brief Title: Vessel Resection and Reconstruction of Biliary Tract Cancers
Status: Completed | Type: Observational
Sponsor: Kansai Hepatobiliary Oncology Group (Network)
Responsible Party: Sponsor
Other Study IDs: KHBO1205; UMIN000010415 (Registry Identifier: UMIN)
Record Dates: First submitted 2013-05-14; First posted 2013-05-23 (Estimated); Last update posted 2014-07-01 (Estimated); Status verified 2014-06

CONDITIONS: Biliary Tract Cancer
MeSH Terms: conditions — Biliary Tract Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
To investigate the vessel resection and reconstruction in biliary tract cancer.

DETAILED DESCRIPTION:
The vessel resection and reconstruction of hepatic artery and portal vein in biliary tract cancer surgery is still controversial. In this study, we retrospectively evaluate the diagnostic image, pathology, peri-operative events, recurrence, and prognosis in these patients, as a multi-center surveillance.

ELIGIBILITY:
Inclusion Criteria:

* Cases of vessel resection and reconstruction in biliary tract cancer.

Exclusion Criteria:

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients who underwent vessel resection and reconstruction in biliary tract cancer after 1990 will be included for analysis.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2013-03; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Comparison of vascular invasion in diagnostic image and in pathology. | 20 years
R0 resection rate | 20 years

CONTACTS AND LOCATIONS:
Overall Officials: Hiroaki Nagano, MD, PhD, Study Director — Osaka University Graduate School of Medicine
Locations (1):
- Osaka University, Graduate School of Medicine, Osaka, Osaka, Japan